CLINICAL TRIAL: NCT05862493
Title: Preoperative Focused Cardiac Ultrasound in Hip Fracture Surgery - Study Protocol for a Randomized Controlled Trial
Brief Title: Preoperative Focused Cardiac Ultrasound in Hip Fracture Surgery (PrEcho)
Acronym: PrEcho
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dnr 2022-05628-01
Record Dates: First submitted 2023-04-27; First posted 2023-05-17 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Echocardiography; Hip Fractures; Risk Assessment; Anesthesia; Hemodynamic Instability
Keywords: FOCUS; Point-of-care echocardiography
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: This is a randomized, open label, superiority trial with a 1:1 allocation ratio
Masking Description: Blinded data analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard management (No Intervention): Standard preoperative management, no preoperative TTE
- FOCUS optimization (Experimental): Standard preoperative management AND preoperative FOCUS along with an individualized hemodynamic optimization based on FOCUS findings.
  Interventions: Diagnostic Test: FOCUS echocardiography

INTERVENTIONS:
Diagnostic Test: FOCUS echocardiography — Preoperative FOCUS echocardiography. Based on FOCUS information: correction of low level of venous return and/or step-up monitoring and/or vasoactive drugs
  Arms: FOCUS optimization

SUMMARY:
The primary objective of this study is to investigate the impact of preoperative focused transthoracic ultrasound (FOCUS) on intraoperative hypotension and postoperative complications in hip fracture surgery. Our hypothesis is that a preoperative FOCUS along with a hemodynamic optimization protocol will reduce the occurrence of intraoperative drops in blood pressure and post-operative complications.

DETAILED DESCRIPTION:
Hip fracture surgery is a common procedure, and despite progress in perioperative management, cardiac complications are common, and the post-operative mortality remains high. In this geriatric patient population, cardiac disease as well as varying degrees of dehydration is common, and preoperative knowledge of these conditions have a key role in enabling a proactive perioperative hemodynamic management. However, clinical assessment is surprisingly unreliable and has been shown to easily fail to identify significant cardiac disease and lack of venous return.

Transthoracic echocardiography (TTE) is a well-established and non-invasive investigation that can identify cardiac disease and aberrations in volume status prior to surgery. In a preoperative practice, the use of focused cardiac ultrasound (FOCUS) enables an individualized anesthesia management and has been demonstrated to influence anesthesiologist decision making. Furthermore, measurements of inferior vena cava used as a surrogate for venous return have been shown to be a predictor of intraoperative hypotension.

Patients scheduled for daytime hip fracture surgery will be screened for eligibility.

Random allocation (1:1 allocation ratio) of patients to receive standard care (control group) or standard care + preoperative focused cardiac ultrasound with a preoperative hemodynamic optimization (intervention group). Registration of pre- and intraoperative blood pressure, as well as post-operative complications and mortality will be conducted.

Primary outcome measure: Intraoperative hemodynamic instability defined as MAP < 60 mmHg.Secondary outcome measures: Time to surgery, length of hospital stay, renal failure, cardiac complications (myocardial ischemia, heart failure, post-operative atrial fibrillation, pulmonary edema, pulmonary embolism), 7-,30- and 90-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 65 years of age, with American Socieity of Anesthesiologists (ASA) physical status classification 2-4, that are scheduled for acute hip fracture surgery (ICD-codes s72.0, s72.00, s72.01, s72.1, s72.2)

Exclusion Criteria:

* Metastatic cancer and/or suspect pathological fracture.
* Concurrent other fracture/surgery.
* Reoperation within 72 hours from primary operation.
* Severe dementia.
* Preoperative echocardiography for other reason than participation in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure drop | From date of randomization up to 4 hours
  Intraoperative drop in blood pressure defined as mean arterial pressure (MAP) < 60 mmHg

SECONDARY OUTCOMES:
Change of blood pressure level | From date of randomization up to 4 hours
  Blood pressure (MAP) change from baseline BP
Lowest level of blood pressure (MAP) | From date of randomization up to 4 hours
  Absolut lowest blood pressure (MAP) from baseline BP
Acute kidney failure | From date of randomization up to 48 hours
  Acute kidney damage defined as a raise in serum creatinine according to the KDIGO-criteria
Myocardial injury | From date of randomization up to 48 hours
  Myocardial injury defined as a raise in serum high-sensitive troponin with at least 5 ng/l-1 to a minimum concentration of at least 20 ng/l-1
Readmission | From date of randomization up to 7 days
  Readmission to hospital within 7 days
Mortality | From date of randomization up to 90 days
  Postoperative mortality at 7-, 30- and 90-days

CONTACTS AND LOCATIONS:
Overall Officials: Tomi P Myrberg, MD, PhD, Principal Investigator — Umeå University

IPD SHARING:
Plan to Share IPD: No
SPSS data file will be available for a reasonable request